CLINICAL TRIAL: NCT03789565
Title: Gingival Crevicular Fluid and Serum Levels of Hepcidin, IL-6 and IL-10 in Periodontal Health and Disease
Brief Title: Hepcidin Levels in Periodontal Health and Disease
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, ÇİĞDEM COŞKUN TÜRER, clinical associate professor, DDS, PhD, Bulent Ecevit University
Other Study IDs: hepcidin
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Periodontal Diseases
Keywords: periodontal diseases; hepcidin; elisa; interleukin 6; interleukin 10
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid and Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1. Healthy individuals from periodontal perspective:: GI < 1, PD ≤ 3 mm, CAL = 0 mm, with no apparent bone loss on radiography.
  Interventions: Other: Biomarker test
- Group 2. Individuals diagnosed with Gingivitis: GI > 1, PD ≤ 3 mm, CAL = 0 mm, with no apparent bone loss on radiography.
  Interventions: Other: Biomarker test
- Group 3. Individuals diagnosed with CP: GI > 1, PD ≥ 5 mm, CAL ≥ 3 mm, with apparent bone loss on radiography.
  Interventions: Other: Biomarker test

INTERVENTIONS:
Other: Biomarker test — Diagnostic biomarker study

SUMMARY:
Periodontal disease refers to inflammatory disease of the periodontium caused by the host and/or pathogenic microorganisms. Anti-inflammatory and pro-inflammatory cytokines play a role in the periodontal inflammation process. The aim of this study was to evaluate the levels of hepcidin, interleukin (IL)-6, and IL-10 levels in gingival crevicular fluid (GCF) and in serum samples obtained from individuals with periodontal inflammation.

DETAILED DESCRIPTION:
The study included 90 individuals, who were divided into three groups: periodontally healthy (PH) (n=30); gingivitis (G) (n=30); and chronic periodontitis (CP) (n=30). GCF and serum samples were obtained from each individual, and samples were evaluated using ELISA. Statistical evaluation of the data was performed using the SPSS packet data program.

ELIGIBILITY:
Inclusion Criteria:

* Systematically healthy patients. Patients who did not receive any medication or periodontal treatment within the previous 6 months

Exclusion Criteria:

* Individuals who smoked and women who were pregnant and/or lactating were excluded from the study

Ages: 32 Years to 52 Years | Sex: All
Age Groups: Adult
Study Population: The study included a total of 60 individuals between 32 and 52 years of age, with a total number of teeth > 20, who underwent consultation for periodontal treatment
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Hepcidin levels | 1 year
  Change in inflammatory phases

SECONDARY OUTCOMES:
IL-6 levels | 1 year
  Change in inflammatory phases
IL-10 levels | 1 year
  Change in inflammatory phases

CONTACTS AND LOCATIONS:
Locations (1):
- Çiğdem Coşkun Türer, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No